CLINICAL TRIAL: NCT02674490
Title: Effects of Transcranial Direct Current Stimulation (tDCS) Plus Language Therapy for Naming in Subacute Left Hemisphere Stroke
Brief Title: Stimulating Language in Subacute StrokE
Acronym: SLISSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00089018
Record Dates: First submitted 2016-01-27; First posted 2016-02-04 (Estimated); Results first posted 2022-09-30 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Stroke
Keywords: aphasia, language
MeSH Terms: conditions — Stroke; Aphasia; Language | interventions — Transcranial Direct Current Stimulation; Salts

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A-tDCS & SALT (Experimental): A-tDCS (1 mA) plus Speech and Language Treatment (SALT) for 15 sessions (20-minutes per each 45-minute treatment session) over the course of 3 weeks. The electrical current will be administered to a pre-specified region of the brain. The stimulation will be delivered at an intensity of 1mA for a maximum of 20 minutes. SALT will be a computer-delivered naming + picture matching task .
  Interventions: Device: A-tDCS (1 mA); Behavioral: SALT
- Sham-tDCS & SALT (Sham Comparator): Sham-tDCS plus SALT for 15 sessions (20-minutes per each 45-minute treatment session) over the course of 3 weeks. Current will be administered in a ramp-like fashion, but after the ramping, the intensity will drop to 0 mA. SALT will be a computer delivered oral naming + picture naming task.
  Interventions: Behavioral: SALT; Device: Sham

INTERVENTIONS:
Device: A-tDCS (1 mA) — 1 mA of A-tDCS stimulation is induced between two 5 cm x 5 cm saline soaked sponges where one sponge (anode: A-tDCS) is placed on the scalp over the targeted cortical region. Ramping up of the current to 1 mA occurs over 10-15 seconds to allow participants to habituate to the tingling sensation. A-tDCS stimulation will be active only in the first 20 minutes of the 45-minute treatment session.
  Other Names: Anodal transcranial direct current stimulation
  Arms: A-tDCS & SALT
Behavioral: SALT — Computer-delivered naming treatment requires matching word (heard and seen being produced by the speaker) with pictures depicting common objects. It is run on a laptop computer with headphones and 2 large response buttons. During treatment, a picture appears on the laptop screen for 2 seconds. Then, a video of the speaker's face below the nose is presented on the screen saying a word that either matches or does not match the picture. The participant is instructed to press a green response button if the word matches the picture and press the red response button if the word does not match the picture.
  Other Names: Speech and Language Treatment
Device: Sham — 1 mA of A-tDCS stimulation is induced between two 5 cm x 5 cm saline soaked sponges where one sponge (anode: A-tDCS) is placed on the scalp over the targeted cortical region. Ramping up of the current to 1 mA occurs over 10-15 seconds to allow participants to habituate to the tingling sensation. Then, the current will be ramped back down to 0 mA in the sham condition. Termination of the stimulation after the ramping up process is generally undetectable, and the brief duration of stimulation yields no functional effects.
  Other Names: Sham-tDCS
  Arms: Sham-tDCS & SALT

SUMMARY:
The investigators will study the effects of transcranial direct current (tDCS) stimulation during language therapy for naming in individuals with aphasia in the acute and subacute post stroke period. Naming difficulties are a persistent and common symptom in aphasia after left-hemisphere (LH) stroke. Behavioral therapy (speech and language therapy; SALT) is the mainstay treatment for post stroke aphasia. Transcranial direct cortical stimulation (tDCS) is a promising adjunct to traditional SALT. tDCS is a safe, non-invasive, non-painful electrical stimulation of the brain which modulates cortical excitability by application of weak electrical currents in the form of direct current brain polarization. It is usually administered via saline-soaked surface sponge electrodes attached to the scalp and connected to a direct current stimulator with low intensities. Most studies are conducted in the chronic phase after stroke. Because neuroplasticity is greatest early after stroke, there is reason to believe tDCS might be most effective in the acute-subacute period. However, only two studies have evaluated tDCS paired with language therapy in group studies of acute to subacute aphasic stroke patients and only one of these was sham-controlled. Furthermore, no studies (of which we are aware) have combined tDCS with therapy to facilitate naming in post stroke aphasia, as shown to be effective in studies of chronic stroke. In this study, the investigators will evaluate whether tDCS combined with SALT improves naming in individuals with aphasia in the acute and subacute post stroke period, more than SALT alone in a randomized, double-blind, sham-controlled trial. The investigators will test the hypothesis that anodal tDCS (A-tDCS) over a targeted region and computer-delivered SALT is associated with greater gains in accuracy in naming pictures, compared to sham combined with the same computer-delivered SALT in post stroke aphasia.

DETAILED DESCRIPTION:
After informed consent is received, a neurological examination will be performed and multiple screening assessments will be conducted including a tDCS and MRI safety screening. If the participant passes the initial screening portion, speech and language diagnostic testing will be conducted during the same visit (Visit 1). During the next visit (Visit 2), participants will undergo a second baseline assessment of naming ability and assessment of connected speech. On that visit, participants who have no contraindication for MRI (and agree to have MRI) will be randomized to (1) functional magnetic resonance (fMRI) electrode placement or (2) structural electrode placement. All participants who have no contraindication will have structural and resting state functional connectivity MRI (rsfcMRI). Those randomized to fMRI electrode placement will also participate in the naming paradigm during the MRI. The third visit will include electrode positioning and tDCS treatment administration. Participants will receive 15 sessions (Visits 3-17) of tDCS + SALT administration. At the beginning of Visit 3, eligible participants will be randomized to receive either A-tDCS (1 milli amp (mA)) or sham-tDCS (placebo) for 15 sessions (20-minutes per each 45-minute behavioral treatment session) over the course of three weeks. A computer-delivered naming treatment will be coupled with the stimulation. The computer-delivered treatment task will be 45-minutes in total length, so that it will commence at the same time as the tDCS administration and continue for another 25-minutes after the tDCS has ceased. To assess cardiovascular arousal, blood pressure and heart rate will be measured before and after each session. Additionally, discomfort ratings will be recorded following the end of each session using the Wong-Baker FACES Pain Rating Scale and a weekly neurological exam will be administered by a neurologist. Neither the participant nor the clinician monitoring and setting up the treatment will have knowledge of the treatment condition (A-tDCS versus sham). Utilizing a computerized picture naming assessment, all participants will be assessed at several different time points throughout the experiment: twice immediately before and twice the week immediately following the fifteenth and final treatment session; twice at five weeks follow-up after the end of treatment; and twice at 20 weeks after the end of treatment. Participants who agree to participate in the MRI portion of the study (and have none of the additional exclusion criteria for MRI) will have structural and rsfcMRI at Visit 2, following the 15th treatment session (Week 1 after the end of treatment), and at 5 weeks after the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participant Inclusion Criteria

Participants must satisfy the following inclusion criteria to be considered eligible for entry into this study:

1. Participants must have sustained an acute ischemic left hemisphere stroke.
2. Participants must be fluent speakers of English by self-report.
3. Participants must be capable of giving informed consent or indicating another to provide informed consent.
4. Participants must be age 18 or older.
5. Participants must be premorbidly right handed.
6. Participants must be within 3 months of onset of stroke.
7. Participants must have an aphasia diagnosis as confirmed by the Western Aphasia Battery-Revised.
8. Participants must achieve at least 65% accuracy on screening task (comparable to treatment task) on 1 of 3 attempts

Exclusion Criteria:

* Participant Exclusion Criteria

Participants with any of the following characteristics will not be eligible for entry into this study:

1. Previous neurological or psychiatric disease, including previous symptomatic stroke.
2. Seizures during the previous 12 months.
3. Uncorrected visual loss or hearing loss by self-report.
4. Use of medications that lower the seizure threshold (e.g., methylphenidate, amphetamine salts).
5. Use of N-methyl-D-aspartate (NMDA) antagonists (e.g., memantine).
6. History of brain surgery or any metal in the head.
7. Scalp sensitivity (per participant report).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2016-06-15 (Actual); Primary Completion 2021-11-12 (Actual); Study Completion 2022-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Argye B Hillis-Trupe, MD, MA, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon completion of the projects and dissemination of primary study results, the analysis data files will be made available to the public, along with the final version of the study protocol, the data dictionary, and brief instructions ("Read me" file). The public use data files and the accompanying documents will be made available through the National Technical Information Service (NTIS).

REFERENCES:
- [Derived] Kang JS, Bunker LD, Stockbridge MD, Hillis AE. White Matter Hyperintensities as a Predictor of Aphasia Recovery. Arch Phys Med Rehabil. 2024 Jun;105(6):1089-1098. doi: 10.1016/j.apmr.2024.01.008. Epub 2024 Jan 26. PMID 38281579
- [Derived] Stockbridge MD, Elm J, Teklehaimanot AA, Cassarly C, Spell LA, Fridriksson J, Hillis AE. Individual Differences in Response to Transcranial Direct Current Stimulation With Language Therapy in Subacute Stroke. Neurorehabil Neural Repair. 2023 Aug;37(8):519-529. doi: 10.1177/15459683231190642. Epub 2023 Aug 17. PMID 37592860
- [Derived] Stockbridge MD, Elm J, Breining BL, Tippett DC, Sebastian R, Cassarly C, Teklehaimanot A, Spell LA, Sheppard SM, Vitti E, Ruch K, Goldberg EB, Kelly C, Keator LM, Fridriksson J, Hillis AE. Transcranial Direct-Current Stimulation in Subacute Aphasia: A Randomized Controlled Trial. Stroke. 2023 Apr;54(4):912-920. doi: 10.1161/STROKEAHA.122.041557. Epub 2023 Mar 13. PMID 36912144

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | A-tDCS & SALT | Sham-tDCS & SALT
Started (Randomized) | 30 | 28
Received at Least One Treatment Session (Modified Intent-to-treat Sample) | 26 | 25
Completed (Completed 1 week follow-up) | 25 | 21
Not Completed | 5 | 7

BASELINE CHARACTERISTICS:
Population: The primary analysis was conducted for the modified Intent-to-treat sample defined as all randomized participants for whom study treatment was initiated.
Groups:
- Total: Total of all reporting groups
Arm/Group | A-tDCS & SALT | Sham-tDCS & SALT | Total
Number analyzed (Participants) | 26 | 25 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.1 (12.2) | 63.8 (15) | 64.5 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 14 | 24
  Male | 16 | 11 | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Participants could indicate multiple race/ethnicities
  Participants
    White | 19 | 13 | 32
    Black | 6 | 10 | 16
    Other/Unknown | 1 | 2 | 3
    Hispanic | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26 | 25 | 51
Western Aphasia Battery Aphasia Quotient [Median (Inter-Quartile Range); unit: units on a scale] — The scores range from 0-100. Higher scores are associated with better language.
  units on a scale | 68.9 [47.9 to 87.0] | 59.9 [33.5 to 82.3] | 66.1 [40.9 to 85.7]
NIH Stroke Scale [Median (Inter-Quartile Range); unit: units on a scale] — The scale ranges from 0-42 with lower scores being better. A score of 0 indicates no stroke symptoms. A score of 42 indicates severe stroke.
  units on a scale | 2 [2 to 3] | 5 [4 to 9] | 4 [2 to 6.5]

OUTCOME MEASURES:

1. Primary Outcome: Change in Accuracy of Naming Untrained Pictures (Philadelphia Naming Test (PNT)) Pre-treatment to 1 Week Post-treatment
Description: The purpose of this measure was to determine whether A-tDCS coupled with SALT will improve naming performance of participants with post stroke aphasia more effectively than SALT alone (i.e., the sham condition).
  The PNT is a 175-item picture naming test where a person earns one point per each correct answer. Scores range from 0-175 with higher scores associated with better performance.
  The outcome measure was the difference between the average of administrations on two consecutive days immediately before treatment and administrations on two consecutive days within 1 week after the end of treatment.
Time Frame: 2 consecutive days immediately before treatment and 2 consecutive days within 1 week after the end of treatment
Population: The mITT=modified Intent-to-treat sample is defined as all randomized participants for whom study treatment was initiated (e.g. attended at least one treatment session), regardless of the treatment actually received. Participants were analyzed according to the group to which they were randomized. Missing data was imputed using multiple imputation. The primary analysis was adjusted for aphasia type (Anomia, Broca, or other type), baseline aphasia severity (AQ), and age.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | A-tDCS & SALT | Sham-tDCS & SALT
Number analyzed (Participants) | 26 | 25
score on a scale | 22.3 [13.5 to 31.2] | 18.5 [9.6 to 27.4]
Statistical Analysis 1: Comparison: A-tDCS & SALT vs Sham-tDCS & SALT; Sample Size Determination If sample size in each group is 20, we will have 89% power to detect a difference in means of 23 (the difference between A-tDCS mean change in accuracy of 33 and a sham mean change in accuracy of 10) assuming that the SD of change for both groups is 22.2 using a two group t-test with a two-sided alpha of 0.05; Test type: Superiority; p = 0.54, Regression, Linear — Threshold for significance is two-sided alpha of 0.05; The primary analysis was adjusted for aphasia type (Anomia, Broca, or other type), baseline aphasia severity (AQ), and age

2. Secondary Outcome: Change in Accuracy of Naming Untrained Pictures (Philadelphia Naming Test) Pre-treatment to 5-weeks Post-treatment
Description: To determine whether A-tDCS coupled with SALT will improve naming performance of participants with post stroke aphasia for a greater duration than SALT alone (i.e., the sham condition). The PNT is a 175-item picture naming test where a person earns one point per each correct answer. Scores range from 0-175 with higher scores associated with better performance.
Time Frame: The PNT will be administered at baseline and at 5 weeks post treatment.
Population: Completers sample. Missing data is not imputed. Data was missing for 6 participants.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | A-tDCS & SALT | Sham-tDCS & SALT
Number analyzed (Participants) | 25 | 20
score on a scale | 29.95 [18.84 to 41.07] | 20.82 [9.36 to 32.27]

3. Secondary Outcome: Change in Content of Picture Description Pre-treatment to 1 Week Post-treatment
Description: The investigators will also record the description of the "Cookie Theft" picture during administration of the National Institutes of Health Stroke Scale before and after treatment, and count the number of Content Units (CU) mentioned by healthy controls. This measure provides a sensitive measure of content of narrative speech in all levels of aphasia.
  Content Units are previously identified aspects of a picture that describe what is portrayed. The Cookie Theft picture includes 30 CUs on the left and 23 on the right combined into a single measure (the total). A person earns one point per each piece of content included. Scores range from 0-53 with higher scores associated with better performance.
Time Frame: Immediately before and within 1 week after treatment
Population: Completers sample. Missing data is not imputed. The data was missing for 9 patients.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | A-tDCS & SALT | Sham-tDCS & SALT
Number analyzed (Participants) | 25 | 17
units on a scale | 4.10 [1.93 to 6.27] | 1.66 [-0.89 to 4.21]

4. Secondary Outcome: Change in Efficiency of Picture Description Pre-treatment to 1 Week Post-treatment
Description: The investigators determined the number of syllables/content unit (CU) in the Cookie Theft description, then calculated the difference between this performance pre-treatment and 1-week post-treatment. Syllables/CU provides a sensitive measure of efficiency of narrative speech in all levels of aphasia. Greater efficiency (fewer syllables required to convey a given amount of content) is associated with improvement in language.
  Content Units are previously identified aspects of a picture that describe what is portrayed. The Cookie Theft picture includes 30 CUs on the left and 23 on the right combined into a single measure (the total). A person earns one point per each piece of content included. Scores range from 0-53 with higher scores associated with better performance.
  A person who does not produce any language would have zero syllables, but there is no maximum number of syllables a person is allowed to produce in response to the task.
Time Frame: Immediately before and within 1 week after treatment
Population: Completers sample. Missing data is not imputed. The data was missing for 9 patients.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | A-tDCS & SALT | Sham-tDCS & SALT
Number analyzed (Participants) | 25 | 17
units on a scale | -12.23 [-19.99 to -4.46] | -1.29 [-11.42 to 8.83]

5. Secondary Outcome: Change in Content of Picture Description Pre-treatment to 5 Weeks Post-treatment
Description: The investigators will also record the description of the "Cookie Theft" picture during administration of the National Institutes of Health Stroke Scale before and after treatment, and count the number of Content Units (CU) mentioned by healthy controls.
  Content Units are previously identified aspects of a picture that describe what is portrayed. The Cookie Theft picture includes 30 CUs on the left and 23 on the right combined into a single measure (the total). A person earns one point per each piece of content included. Scores range from 0-53 with higher scores associated with better performance.
Time Frame: Immediately before and at 5 weeks after treatment
Population: Completers sample. Missing data is not imputed. The data was missing for 10 patients.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | A-tDCS & SALT | Sham-tDCS & SALT
Number analyzed (Participants) | 24 | 17
units on a scale | 5.42 [3.22 to 7.62] | 1.42 [-1.14 to 3.97]

6. Secondary Outcome: Change in Efficiency of Picture Description Pre-treatment to 5 Weeks Post-treatment
Description: The investigators determined the number of syllables/content unit (CU) in the Cookie Theft description, then calculated the difference between this performance pre-treatment and 5-weeks post-treatment. Syllables/CU provides a sensitive measure of efficiency of narrative speech in all levels of aphasia. Greater efficiency (fewer syllables required to convey a given amount of content) is associated with improvement in language.
  Content Units are previously identified aspects of a picture that describe what is portrayed. The Cookie Theft picture includes 30 CUs on the left and 23 on the right combined into a single measure (the total). A person earns one point per each piece of content included. Scores range from 0-53 with higher scores associated with better performance.
  A person who does not produce any language would have zero syllables, but there is no maximum number of syllables a person is allowed to produce in response to the task.
Time Frame: Immediately before and at 5 weeks after treatment
Population: Completers sample. Missing data is not imputed. The data was missing for 10 patients.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | A-tDCS & SALT | Sham-tDCS & SALT
Number analyzed (Participants) | 24 | 17
units on a scale | -12.64 [-20.46 to -4.82] | 2.47 [-7.48 to 12.43]

7. Secondary Outcome: Change in Stroke Impact Scale (SIS) Pre-treatment to Post-treatment
Description: The SIS will be administered at baseline and within 1 week after treatment to evaluate changes in quality of life and social engagement.
  The SIS includes 59 aspects of post-stroke functioning. Participants rate each of the items on a scale from 5 (least encumbered, affected, or difficult) to 1 (most encumbered, affected or difficult). Ratings on each aspect are summed and then transformed to a 100-point scale using the following formula:
  Score = [(Actual raw score - lowest possible raw score) / Possible raw score range] x 100
  The last item (#60) assesses the participant's overall perception of recovery and is presented in the form of a visual analog scale from 0 to 100, where 0 = "no recovery" and 100 = "full recovery."
  Total score is the average of all transformed scores and the overall perception of recovery. Total scores range from 0-100, with higher scores associated with better recovery.
Time Frame: Immediately before and within 1 week after treatment
Population: Completers sample. Missing data is not imputed. The data was missing for 9 patients.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | A-tDCS & SALT | Sham-tDCS & SALT
Number analyzed (Participants) | 22 | 20
units on a scale | 2.56 [-0.72 to 5.83] | 3.85 [0.50 to 7.20]

8. Secondary Outcome: Change in Stroke Impact Scale (SIS) Pre-treatment to 5 Weeks Post-treatment
Description: The SIS was administered at baseline and 5 weeks after treatment to evaluate any lasting changes in quality of life and social engagement.
  The SIS includes 59 aspects of post-stroke functioning. Participants rate each of the items on a scale from 5 (least encumbered, affected, or difficult) to 1 (most encumbered, affected or difficult). Ratings on each aspect are summed and then transformed to a 100-point scale using the following formula:
  Score = [(Actual raw score - lowest possible raw score) / Possible raw score range] x 100
  The last item (#60) assesses the participant's overall perception of recovery and is presented in the form of a visual analog scale from 0 to 100, where 0 = "no recovery" and 100 = "full recovery."
  Total score is the average of all transformed scores and the overall perception of recovery. Total scores range from 0-100, with higher scores associated with better recovery.
Time Frame: Immediately before and 5 weeks after treatment
Population: Completers sample. Missing data is not imputed. The data was missing for 10 patients.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | A-tDCS & SALT | Sham-tDCS & SALT
Number analyzed (Participants) | 23 | 18
units on a scale | 2.08 [-1.17 to 5.33] | 4.18 [0.78 to 7.58]

9. Secondary Outcome: Change in Accuracy of Naming Untrained Pictures (Philadelphia Naming Test) Pre-treatment to 20-weeks Post-treatment
Description: as for outcome 2
Time Frame: The PNT will be administered at baseline and at 20 weeks post treatment.
Population: Completers sample. Missing data is not imputed. The data was missing for 6 patients.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | A-tDCS & SALT | Sham-tDCS & SALT
Number analyzed (Participants) | 24 | 21
score on a scale | 34.04 [22.90 to 45.18] | 25.55 [14.13 to 36.97]

10. Secondary Outcome: Change in Content of Picture Description Pre-treatment to 20-weeks Post-treatment
Description: as for outcome 5
Time Frame: Immediately before and at 20 weeks after treatment
Population: Completers sample. Missing data is not imputed. The data was missing for 10 patients.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | A-tDCS & SALT | Sham-tDCS & SALT
Number analyzed (Participants) | 24 | 17
units on a scale | 5.15 [2.94 to 7.35] | 3.28 [0.72 to 5.85]

11. Secondary Outcome: Change in the Efficiency of Picture Description Pre-treatment to 20 Weeks Post-treatment
Description: The investigators determined the number of syllables/content unit (CU) in the Cookie Theft description, then calculated the difference between this performance pre-treatment and 20-weeks post-treatment. Syllables/CU provides a sensitive measure of efficiency of narrative speech in all levels of aphasia. Greater efficiency (fewer syllables required to convey a given amount of content) is associated with improvement in language.
  Content Units are previously identified aspects of a picture that describe what is portrayed. The Cookie Theft picture includes 30 CUs on the left and 23 on the right combined into a single measure (the total). A person earns one point per each piece of content included. Scores range from 0-53 with higher scores associated with better performance.
  A person who does not produce any language would have zero syllables, but there is no maximum number of syllables a person is allowed to produce in response to the task.
Time Frame: Immediately before and at 20 weeks after treatment
Population: Completers sample. Missing data is not imputed. The data was missing for 10 patients.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | A-tDCS & SALT | Sham-tDCS & SALT
Number analyzed (Participants) | 24 | 17
units on a scale | -14.75 [-22.58 to -6.91] | 6.53 [-3.63 to 16.69]

12. Secondary Outcome: Change in Stroke Impact Scale (SIS) Pre-treatment to 20 Weeks Post-treatment
Description: The SIS was administered at baseline and 20 weeks after treatment to evaluate any lasting changes in quality of life and social engagement.
  The SIS includes 59 aspects of post-stroke functioning. Participants rate each of the items on a scale from 5 (least encumbered, affected, or difficult) to 1 (most encumbered, affected or difficult). Ratings on each aspect are summed and then transformed to a 100-point scale using the following formula:
  Score = [(Actual raw score - lowest possible raw score) / Possible raw score range] x 100
  The last item (#60) assesses the participant's overall perception of recovery and is presented in the form of a visual analog scale from 0 to 100, where 0 = "no recovery" and 100 = "full recovery."
  Total score is the average of all transformed scores and the overall perception of recovery. Total scores range from 0-100, with higher scores associated with better recovery.
Time Frame: Immediately before and 20 weeks after treatment
Population: Completers sample. Missing data is not imputed. The data was missing for 10 patients.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | A-tDCS & SALT | Sham-tDCS & SALT
Number analyzed (Participants) | 23 | 18
score on a scale | 2.60 [-0.65 to 5.86] | 4.28 [0.88 to 7.69]

ADVERSE EVENTS:
Time Frame: 20 weeks
Arm/Group | A-tDCS & SALT | Sham-tDCS & SALT
All-Cause Mortality (participants affected / at risk) | 1/26 | 0/25
Serious Adverse Events (participants affected / at risk) | 2/26 | 2/25
Other Adverse Events (participants affected / at risk) | 5/26 | 1/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A-tDCS & SALT (N=26) | Sham-tDCS & SALT (N=25)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A-tDCS & SALT (N=26) | Sham-tDCS & SALT (N=25)
Application site irritation (General disorders) | 3 (3) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-03-02): https://cdn.clinicaltrials.gov/large-docs/90/NCT02674490/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-18): https://cdn.clinicaltrials.gov/large-docs/90/NCT02674490/SAP_001.pdf
  • Informed Consent Form (2019-11-14): https://cdn.clinicaltrials.gov/large-docs/90/NCT02674490/ICF_002.pdf